CLINICAL TRIAL: NCT03622021
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Dose-Escalation First-In-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AK111 in Healthy Subjects
Brief Title: A Study of AK111 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AK111-101
Record Dates: First submitted 2018-07-27; First posted 2018-08-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- AK111 30mg (Experimental): Single dose of 30mg AK111 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: AK111 or Placebo
- AK111 75mg (Experimental): Single dose of 75mg AK111 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: AK111 or Placebo
- AK111 150mg (Experimental): Single dose of 150mg AK111 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: AK111 or Placebo
- AK111 300mg (Experimental): Single dose of 300mg AK111 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: AK111 or Placebo
- AK111 450mg (Experimental): Single dose of 450mg AK111 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: AK111 or Placebo
- AK111 600mg (Experimental): Single dose of 600mg AK111 or placebo is administered subcutaneously to healthy subjects
  Interventions: Drug: AK111 or Placebo

INTERVENTIONS:
Drug: AK111 or Placebo — All the subjects in each cohort will be randomized in a 3:1 ratio to receive either AK111 or Placebo.

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single dose-escalation first-in human study to evaluate the safety, tolerability, PK, PD and immunogenicity of AK111 in healthy subjects following SC administration. The study will consist of cohorts of healthy subjects. Cohort 1, four unique subjects will be randomized to receive either active AK111 (N=3) or matching placebo (N=1). Cohorts 2, 3, 4 and 5, eight unique subjects will be randomized to receive either active AK111 (N=6) or matching placebo (N=2). Approximately 36 subjects will be treated in this study.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria (as applicable) to be eligible for participation in this study.

1. Have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures.
2. Female or male between 18 and 55 years of age, inclusive, at screening.
3. Must have a calculated body mass index (BMI) 19 ≤ BMI ≤ 32(inclusive) at screening, and a total body weight ≥ 50 kg for male or ≥ 45 kg for female at screening.
4. Females of child bearing potential must have a negative pregnancy test in serum at screening and a negative serum pregnancy test on Day -1, either be of non-child bearing potential, defined as being:

   1. Postmenopausal (for at least 2 years before screening), verified by serum follicle stimulating hormone (FSH) level >40 mIU/mL at screening, or
   2. Permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy), or
   3. Congenitally sterile
5. Women of child-bearing potential must use one of the following methods of contraception, from screening until at least 120 days after dosing:

   A highly effective method with a failure rate of less than 1%:
   * Implant contraceptive (e.g. Jadelle)
   * Intra-uterine device (IUD) containing either copper or levonorgestrel (e.g. Mirena)
   * Male sterilization (vasectomy)
   * Female sterilization (e.g. by bilateral tubal ligation ('tying tubes') or hysterectomy)

   A method for which the failure rate is between 5% and 10% in real life use, in combination with a barrier method (male condom):
   * Injectable contraceptive (e.g. Depo Provera)
   * Oral Contraceptive Pill (combined hormonal pill or progestogen-only 'mini-pill')
   * Vaginal contraceptive ring (e.g. NuvaRing) Please note that condoms alone are not highly effective methods of contraception. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
6. Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use an effective method of contraception as listed above from Day 1 through 120 days after receipt of the last dose of study medication. It is strongly recommended for the female partner of a male subject to also us an effective method of contraception throughout this period.
7. Must, in the opinion of the Investigator, be in good general health based upon medical history, physical examination (including vital signs), 12-lead ECG and clinical laboratory tests must fall within the clinical laboratory's reference normal ranges unless the results have been determined by the Investigator to have no clinical significance).
8. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures as specified in the protocol.

Exclusion Criteria Subjects who meet any of the following exclusion criteria will not be enrolled in this study.

1. Subjects who are investigational site staff members or subjects who are Sponsor employees directly involved in the conduct of the study.
2. Are pregnant, nursing, or planning pregnancy within 120 days following the last dose of study medication (both men and women) while enrolled in the study.
3. Have previously participated in an investigational trial involving administration of any investigational compound within 3 months or 5 half-lives (whichever is longer) prior to the study dosing, or currently participating in another clinical study.
4. Have a planned surgical intervention for a pretreatment condition within the duration of the trial, including the follow up period.
5. Have used any biologic within the previous 12 months prior to the study dosing.
6. Use of any of the following, unless agreed as non-clinically relevant by the Investigator: Prescription medication within 4 weeks prior to the study dosing; Over-the-counter medication (excluding paracetamol) within 7 days prior to the study dosing. Paracetamol use must be limited to 2 g per day and no more than 3 days usage in the 4 weeks prior to the study dosing; Vitamin therapy or dietary supplements within 7 days prior to the study dosing and for the duration of the study; Herbal supplements within 4 weeks prior to the study dosing and for the duration of the study. Medications which are known CYP P450 isoenzyme substrates/inducers/inhibitors must be excluded within 4 weeks prior to study dosing and for the duration of the study.
7. Current acute infection or history of acute infection within 7 days prior to receipt of the study drug; additionally, aural temperature that exceeds 37.4°C at Day -1 (baseline).
8. Have had a serious infection, define as requiring intravenous antibiotics or hospitalization within 3 months prior to screening; Have had recurrent or chronic infection, define as ≥ 3 infections requiring anti-microbials over the past 12 months prior to screening.
9. Have a history of latent or active granulomatous infection, including histoplasmosis, candidiasis (clinically significant candidiasis or recurrent candidiasis), or coccidioidomycosis prior to screening, or a history of any other infectious disease within 4 weeks prior to screening that in the opinion of the investigator, affects the subject's ability to participate in the trial.
10. History or complication of tuberculosis, or evidence of latent tuberculosis by QuantiFERON screening. If the QuantiFERON®-TB Gold test is indeterminate, a retest is allowed if results can be obtained. If the retest is also indeterminate, the subject will be excluded from the study. Subjects who have had household contact with a person with active TB are excluded.
11. Positive for hepatitis B surface antigen, hepatitis C antibodies or HIV at screening.
12. Have had a substance abuse (drug or alcohol) problem within the previous 3 years, or a positive urine drug screen at screening.
13. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 100 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.
14. Use of tobacco or nicotine containing products (including e-cigarettes) at any time within six months before screening and for the duration of the study.
15. Have poor venous access and are unable to donate blood.
16. Have donated blood within 90 days prior to the study dosing.
17. Have a history of multiple drug allergies or a known allergy or hypersensitivity to any biologic therapy at screening that is important in the opinion of the Investigator.
18. Have a known allergy or reaction to any component of the AK111 formulation.
19. Have a history of known demyelinating diseases such as multiple sclerosis or optic neuritis.
20. Have a history of lymphoproliferative disease, including lymphoma, or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location, or clinically significant splenomegaly.
21. Have any known malignancy or have a history of malignancy within the previous 5 years (with the exception of a non-melanoma skin cancer that has been treated with no evidence of recurrence).
22. Have a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to the study dosing).
23. Have an implanted defibrillator or pacemaker.
24. 12-lead ECG demonstrating QTc interval > 450 msec corrected using the Fridericia's formula (QTcF) at screening from average of three ECGs obtained (separated by approximately 1-minute intervals) after 5 minutes of supine rest.
25. Blood pressure >140 mmHg (systolic) or > 90 mmHg (diastolic) at screening, following at least 5 minutes of supine rest. If blood pressure (BP) is >140 mmHg (systolic) or >90 mmHg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
26. Have had a live vaccination within 12 weeks prior to the study dosing, or intend to have a live vaccination during the course of the study, or have participated in a vaccine clinical trial within 12 weeks prior to the study dosing.
27. Have any psychiatric or serious or active medical illness which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include renal, cardiac, hematological, hepatic, pulmonary (including chronic asthma), endocrine (eg, diabetes), central nervous, gastrointestinal (including but not limit to Crohn's disease, ulcerative colitis, an ulcer), vascular, metabolic (thyroid disorders, adrenal disease), or immunodeficiency disorders that are clinically significant or requiring treatment.
28. Are believed, by the Investigator, to be inappropriate for study participation for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent AE/SAEs | From baseline through 12 weeks

SECONDARY OUTCOMES:
The endpoint for assessment of PD including the change from baseline in serum IL-17A level and serum cytokines. | From baseline through 12 weeks
Area under the concentration curve (AUC) of AK111 | From baseline through 12 weeks
Maximum observed concentration (Cmax) of AK111 | From baseline through 12 weeks
Number of subjects who develop detectable anti-drug antibodies (ADAs) [ | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Christchurch Clinical Studies Trust (CCST), Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No